CLINICAL TRIAL: NCT04554576
Title: Escoge Salud (Choose Health) Effects and Sustainability of a Chronic Pain Self-Management Program in Middle to Older Age Hispanic Americans
Brief Title: Escoge Salud (Choose Health): a Chronic Pain Self-Management Program in Middle to Older Age Hispanic Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1326143-3
Record Dates: First submitted 2020-01-02; First posted 2020-09-18 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pain
Keywords: Hispanic American; Latino; self-management training; sustainability; health care utilization
MeSH Terms: conditions — Chronic Pain; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: This is a prospective study with a secondary randomization to a remote, nonfrequent provider feedback sustainability intervention. All participants will receive the 6-week self-management intervention and do pre/post evaluations. After the 6-week intervention, half the group will be randomized to a every 6th week for 6 months healthcare provider phone/video visit session and half will be received to no treatment control for 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6-week self-management and remote feedback for 6 months (Experimental): All participants will receive the 6-week self-management program and after, half the group will be randomized to an every 6th week healthcare provider feedback phone or video visit session for 6 months (4 visits over 24 months).
  Interventions: Behavioral: Chronic Disease Self-Management Program (CDSMP) for chronic pain in Spanish; Behavioral: Remote feedback active group
- 6-week self-management and control group for 6 months (Active Comparator): All participants will receive the 6-week self-management program and after, half will be randomized to a 6 month control grup
  Interventions: Behavioral: Chronic Disease Self-Management Program (CDSMP) for chronic pain in Spanish; Behavioral: Remote feedback control group

INTERVENTIONS:
Behavioral: Chronic Disease Self-Management Program (CDSMP) for chronic pain in Spanish — The CDSMP meets for 2.5 hours for 6 weeks. Topics covered are: understanding pain, finding resources, mindfulness, pain science, pacing, exercise, relaxation, communication, sex/intimacy, healthy eating, weight and medication management, making treatment decisions and confronting fears.
  Participants are encouraged to create their own personal health goals and make weekly action plans to meet their personal goals. Each week participants learn new tools and problem-solving techniques to meet their health goals and themes are repeated throughout 6-week period to ensure understanding and integration. Participants are encouraged to problem-solve and ask questions to the group about creating and carrying out their self-management plan.
  The intervention follows the content of the book Programa de Manejo Personal del Dolor Crónico (Living a Healthy Life with Chronic pain)
  Other Names: CDSMP for chronic pain in Spanish
Behavioral: Remote feedback active group — After the 6-week self management program, half the participants will be randomized to an every 6 weeks for 6 months phone or video visit from a health care provider, in Spanish. The phone or video sessions will include: review previous action-plans (goals) and provide support in forming new action-plans (goals)
  Arms: 6-week self-management and remote feedback for 6 months
Behavioral: Remote feedback control group — After the 6-week self-management program, half the participants will be randomized to a control group for 6 months.
  Arms: 6-week self-management and control group for 6 months

SUMMARY:
The purpose of this study is to evaluate patient satisfaction and health status before and after a 6-week established self-management training program for middle to older age Hispanic Americans living with chronic musculoskeletal pain in a large, hospital based urban health maintenance organization. The secondary aim is to evaluate the effects of remote, nonfrequent healthcare provider feedback for 6 months on health care utilization, health status and patient satisfaction.

DETAILED DESCRIPTION:
Managing chronic pain in the US costs approximately $635 billion and half of this expenditure is for joint and arthritis related pain syndromes. Interestingly, compared with non-Hispanic whites (NHWs), Hispanic Americans (HAs) report significantly lower rates of chronic pain with consistently higher levels of pain intensity in both population and clinically based studies. Chronic musculoskeletal pain (CMP) incidence increases with age and the HA aging population is among the fastest growing segments of the US population. Despite reporting more intense pain, HA are less likely to seek medical care versus NHWs for acute and chronic pain. Lack of access, cultural stoicism and an external locust of control are thought to explain why HAs seek care at a reduced rate. Psychological factors play a significant role in pain experience, HAs may employ catastrophic thinking and experience more pain related anxiety which are predictors of exacerbated pain experience. Pain comorbidities may be amenable to treatment with appropriate, culturally sensitive treatment focusing on enhancing self-efficacy to manage the complex array of psychological pain comorbidities. There is a societal impact of undertreating chronic pain in the HA population. While HAs have the lowest rate of short-term sick usage (<1-2 days), they have the highest rate of long-term sick usage (>31 days). This increased long-term time off puts HAs at risk of losing their job if the time off exceeds Family Leave and Medical Act minimums. Lastly, it is well documented, HAs are hesitant to take strong pain medication and there is conflicting evidence surrounding taking over-the-counter medications for pain management. There is a need to provide culturally sensitive, effective chronic pain management treatments for HAs.

There have been 5 well designed studies (n=931) demonstrating efficacy of a trans-created Spanish version of the Chronic Disease Self-Management Program (CDSMP) for HAs with chronic musculoskeletal pain. CDSMP has demonstrated effectiveness in improving pain intensity, self-efficacy (SE) and health behaviors in a community setting . The intervention is a healthcare provider and/or peer led 2.5 hour self-management training session, 1 time per week for 6 weeks taught in a group setting in Spanish. The program is grounded in Bandura's Social Cognitive Theory and uses goal setting and problem solving as corner stones to create a personalized self-management program. Improvements post-intervention in SE predict sustainability of health behaviors and maintenance of improved health status in the long term. Additionally, remote non-frequent health care provider feedback has been associated with maintenance of health behaviors, however this his not been tested in the HA population.

The purpose of this study is to test the feasibility (patient satisfaction and change in health status) after bringing the CDSMP programming to a large urban hospital based medical center that does not currently offer a culturally sensitive, self-management training program in Spanish middle to older age HAs with chronic pain. The secondary aim is to pilot the effectiveness of an every 6th week phone/video visit feedback visit for 24 months on both health status and healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

1. Spanish Speaking
2. Had 1 or 2 outpatient dispense records of NSAIDS between Jan 1 2018 to Dec 31 2018.
3. 5 doctor office visits between 07/01/2017 - 12/31/2018 for any health program.
4. Non-malignant musculoskeletal pain for at least 6 months
5. Interested in learning self-management
6. Ability to have telephone/video visit every 6 weeks
7. Ability to travel to medical center 1x/week for 6 weeks in the afternoon for 2.5 hours

Exclusion Criteria:

1. Major psychiatric or substance abuse problem
2. Mild cognitive impairment/dementia
3. Malignant pain or terminal illness
4. Listed in the Non-contact database

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Self Efficacy | baseline to 6-weeks
  Spanish Arthritis self-efficacy scale (ASES). This tool has 8 questions rating 'certainty' in ability to manage health and chronic pain. It is scored on a visual analogue scale from 1-10, 1= very uncertain to 10= very certain. Higher scores indicate more self-efficacy.
Patient Reported Outcome Measurement Information System (PROMIS) Global Health | baseline to 6-weeks
  Spanish PROMIS Global Health v1.2 measures global physical, mental and social health. It has 10 questions, 9 of which are answered on a 5-point Likert scale and 1 question on a visual analogue scale where 0=no pain and 10=worst pain imaginable. PROMIS measures are scored on a t-score metric where 50 is set to be the population norm and higher scores indicate better global health.
Pain Catastrophizing | baseline to 6-weeks
  Spanish Pain Catastrophizing Scale (PCS) evaluates 3 distinct phenomenon which are characterized by feelings of helplessness, active rumination and excessive magnification associated with pain experience. The questionnaire has 13 questions and is scored on a 5-point Likert scale, 0= not at all to 4 = all the time. Higher scores indicate more catastrophizing.
Health Distress | baseline to 6-weeks
  Health Distress Scale evaluates distress and worry due to illness. It has 4 question that are answered on a 5-point Likert scale where 0= none of the time and 5= all of the time. Higher scores indicate more distress and worry.
Patient Satisfaction | baseline to 6-weeks
  Adapted from Camino con Gusto study. 3 questions on satisfaction with the intervention scored on scored on a 4-point scale: 1 = Strongly disagree, 2 = Disagree, 3 = Agree, 4 = Strongly agree.
Patient Global Impression | baseline to 6-weeks
  Patient Global Impression of Change (PGIC) captures the patients satisfaction with the intervention by asking "How satisfied or dissatisfied are you with the self-management program?' and is scored on a 7-point scale where 7-point scale where -3 =very dissatisfied 0= neither satisfied or dissatisfied and 3= very satisfied.

SECONDARY OUTCOMES:
Doctors office visits | 6 weeks to 30-34 weeks
  Number of Primary Care doctors office visits
Emergency Room use | 6 weeks to 30-34 weeks
  Number of Emergency Room visits
Self Efficacy | 6-weeks to 30-34 weeks
  Spanish Arthritis self-efficacy scale (ASES). This tool has 8 questions rating 'certainty' in ability to manage health and chronic pain. It is scored on a visual analogue scale from 1-10, 1= very uncertain to 10= very certain.
PROMIS Global Health | 6-weeks to 30-34 weeks
  Spanish PROMIS Global Health v1.2 measures global physical, mental and social health. It has 10 questions, 9 of which are answered on a 5-point Likert scale and 1 question on a visual analogue scale where 0=no pain and 10=worst pain imaginable.
Pain Catastrophizing | 6-weeks to 30-34 weeks
  Spanish Pain Catastrophizing Scale (PCS) evaluates 3 distinct phenomenon which are characterized by feelings of helplessness, active rumination and excessive magnification associated with pain experience. The questionnaire has 13 questions and is scored on a 5-point Likert scale, 0= not at all to 4 = all the time
Health Distress | 6-weeks to 30-34 weeks
  Health Distress Scale evaluates distress and worry due to illness. It has 4 question that are answered on a 5-point Likert scale where 0= none of the time and 5= all of the time

CONTACTS AND LOCATIONS:
Overall Officials: Amy Gladin, DPT, Principal Investigator — senior physical therapist
Locations (1):
- KaiserPermanente, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The study will share de-identified health status pre/post and healthcare utilization information to other investigators upon request
Supporting Information: CSR
Time Frame: December 2019 to December 2020
Access Criteria: Available to Investigators upon request